CLINICAL TRIAL: NCT07122999
Title: Effectiveness of Autoinflation on the Recurrence of Otitis Media With Effusion After Tympanostomy Tube Extrusion: A Randomized Controlled Trial
Brief Title: Autoinflation as a Eustachian Tube Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-016-092
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Otitis Media With Effusion (OME); Eustachian Tube Dysfunction
Keywords: Autoinflation; Recurrence; Middle Ear Ventilation; Otitis Media with Effusion
MeSH Terms: conditions — Otitis Media with Effusion; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Autoinflation (Experimental): Participants perform autoinflation using the Eustachi device twice daily for 5 weeks after TT extrusion.
  Interventions: Device: Eustachi
- Observation (No Intervention): Participants are followed without autoinflation after TT extrusion (standard observation only).

INTERVENTIONS:
Device: Eustachi — A handheld device that delivers pulsed air through the nasal passage to facilitate opening of the eustachian tube. Participants in this group use the device twice daily for 5 weeks after tympanostomy tube extrusion.
  Arms: Autoinflation

SUMMARY:
This randomized controlled trial evaluated the effectiveness of autoinflation in preventing recurrence of otitis media with effusion (OME) and reducing the need for reoperation after tympanostomy tube (TT) extrusion in children. Sixty-six pediatric patients with chronic OME underwent TT placement, and 54 were included in the final analysis. After TT extrusion, participants were randomized into two groups: an autoinflation group using a handheld device (Eustachi) for five weeks, and an observation-only group. Patients were followed for two years post-extrusion, with periodic otoscopic and tympanometric assessments.

The autoinflation group showed a lower recurrence rate (19.2%) compared to the observation group (35.7%), although this difference was not statistically significant. However, the reoperation rate was significantly lower in the autoinflation group (7.7% vs. 28.6%). Tympanometric findings suggested more stable middle ear pressure in the autoinflation group. These results indicate that autoinflation is a safe, feasible, and non-invasive method that may support eustachian tube function and reduce the need for repeat TT placement in children following TT extrusion.

DETAILED DESCRIPTION:
Otitis media with effusion (OME) is a prevalent pediatric condition that may lead to hearing loss and developmental delay. Tympanostomy tube (TT) placement is the standard treatment for persistent OME but does not address the underlying cause, and recurrence is common after TT extrusion. This study investigated whether autoinflation after TT extrusion could reduce OME recurrence and the need for reoperation.

In this prospective randomized controlled trial, 66 children aged 3 to 8 years with chronic OME were enrolled at a tertiary hospital. All underwent TT placement under general anesthesia and were followed bi-monthly in the outpatient clinic. After TT extrusion, 54 patients were randomized to either the autoinflation group (n = 26) or the observation group (n = 28). The autoinflation group used the Eustachi device twice daily for five weeks, with instructions provided to children and caregivers. Patients with adenoid hypertrophy, craniofacial anomalies, active otologic disease, or severe systemic disease were excluded.

Outcome measures included OME recurrence and TT reoperation rates over two years, evaluated through otoscopy and tympanometry. The recurrence rate was lower in the autoinflation group (19.2%) than in the observation group (35.7%), though the difference was not statistically significant. However, the reoperation rate was significantly lower in the autoinflation group (7.7%) compared to the observation group (28.6%, p = 0.048). Tympanometry results also showed stable middle ear pressure in the autoinflation group, whereas the observation group experienced a decline in type A tympanograms and an increase in type C patterns over time.

These findings suggest that autoinflation may promote functional rehabilitation of the eustachian tube and maintain middle ear ventilation after TT extrusion. The intervention was well tolerated and feasible in a home setting with caregiver supervision. While autoinflation should not replace TT placement in persistent OME, it may serve as a valuable non-invasive strategy to reduce the risk of recurrence and the need for repeat surgery. Limitations include sample size and lack of quantitative compliance data, warranting future multicenter studies for validation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 8 years
* Clinical diagnosis of chronic otitis media with effusion (OME)
* Underwent tympanostomy tube (TT) placement for persistent OME lasting more than 3 months
* Capable of performing autoinflation, as assessed by the physician
* Caregiver willing to provide informed consent and assist with at-home device use

Exclusion Criteria:

* Presence of adenoid hypertrophy or tonsillar hypertrophy
* History of craniofacial anomalies (e.g., cleft palate)
* Current otologic disease such as otorrhea or tympanic membrane perforation
* Acute otitis media or signs of active inflammation at enrollment
* Underlying severe systemic disease or immunodeficiency
* Inability or refusal to follow autoinflation protocol

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of otitis media with effusion (OME) | Up to 24 months after tympanostomy tube extrusion
  The proportion of patients with a recurrence of OME in the affected ear(s), diagnosed by otoscopy and/or tympanometry, during a 2-year follow-up period after tympanostomy tube extrusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, Seo-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared for this study. This decision was made due to privacy considerations and the absence of a formal data-sharing plan.

REFERENCES:
- [Result] Perera R, Glasziou PP, Heneghan CJ, McLellan J, Williamson I. Autoinflation for hearing loss associated with otitis media with effusion. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD006285. doi: 10.1002/14651858.CD006285.pub2. PMID 23728660